CLINICAL TRIAL: NCT07313449
Title: Study of the Clinical and Radiographic Results of a Fixed Polyethylene Posteriorly Stabilized Cemented Total Knee Prosthesis With a Minimum Follow-up of 1 Year.
Acronym: PTG-Anatomic
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9534
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
Keywords: Osteonecrosis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The knee replacement market is experiencing constant growth. Alongside this growth, there is also an increasing interest in customizing implantation based on specific phenotypes to restore the morphology of the native knee. For example, in the last five years, 2019 publications on knee prosthesis alignment have been identified on PubMed.

It seems worthwhile to study and analyze the performance of the prosthesis used in the Orthopedic Surgery Department of the Strasbourg University Hospitals (HUS) and to compare it with results from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who underwent total knee replacement (TKR) between January 2013 and December 2024
* Patient who underwent an Anatomic, Amplitude, posteriorly stabilized, fixed polyethylene, cemented TKR
* Patient operated on by Professor F. Bonnomet
* Available radiological data: preoperative, immediate postoperative, and postoperative at a minimum of 1 year follow-up

Exclusion Criteria:

- Revision of the arthroplasty during the study follow-up period for a cause not investigated in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient who underwent total knee replacement (TKR) between January 2013 and December 2024
  - Patient who underwent an Anatomic, Amplitude, posteriorly stabilized, fixed polyethylene, cemented TKR
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
IKS / KSS (Knee Society Score) | Up to 12 months
  The classic IKS (often called KSS) has 2 separate scores, each out of 100 points:
  1. Knee Score (Objective / Clinical) - 0 to 100
     Assesses the knee itself:
     * Pain (0-50)
     * Range of motion (0-25)
     * Stability (0-25)
  2. Function Score - 0 to 100
     * Assesses patient function:
     * Walking distance (0-50)
     * Stair climbing (0-50)
  Interpretation (commonly used):
  * 80-100: Excellent
  * 70-79: Good
  * 60-69: Fair
  * < 60: Poor

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique et de Traumatologie du Membre Inférieur - CHU de Strasbourg - France, Strasbourg, France